CLINICAL TRIAL: NCT03327233
Title: Integrated Personalized Connected Care for Complex Chronic Patients - Community-based Management
Brief Title: CONNECARE-Assuta-Case Study 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assuta Medical Center (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Dr Bellaa Azria, Head of Medicine, Assuta Medical Centers, Assuta Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0033-17-ASMC
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Chronic Disease; Old Age; Debility
MeSH Terms: conditions — Chronic Disease; Frailty

STUDY DESIGN:
Intervention Model Description: Matched intervention - control group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implementing the Connecare system to support integrated care for complex patients with an unplanned admission to Assuta Ashdod who are discharged back to the community with an emphasis on Connecare self managment system for the patient and close follow up and coordination of all of the medical, health and social care in the community by a Maccabi integrated care nurse for a period of 3 months post discharge.
  Interventions: Device: Connecare self managment system
- Matched control group (No Intervention): The control group will be selected from Maccabi's database and will be patients who are matched 1:1 with the intervention sample and live in another community similar to Ashdod in socioeconomic characteristics who undergo the same elective major surgery in other hospitals

INTERVENTIONS:
Device: Connecare self managment system — The CONNECARE SMS will rely on a hybrid solution that, besides being autonomous (the patient may use the SMS to monitor and access to her/his data and information), has also a collaborative component (through the interaction with the SACM) to allow participation by clinicians and to provide feedback to them. In so doing, the patient may control her/his activity, receiving recommendations to improve the treatment and to be encouraged in following it.
  Arms: Intervention group

SUMMARY:
The European Union's Horizon 2020 project issued a Call for Action [1] in December 2013 to design, develop, disseminate and evaluate new IT technologies for use in integrative treatment processes, with emphasis on complex adult patient. Assuta Hospital submitted a proposal for this call, as part of a broad consortium of 10 participants from various European countries.

The CONNECARE consortium has formulated a general model for integrative treatment, and is currently in the technological development stages, to create a smart (supportive decision) and adaptive system that supports integrative treatment processes both in the hospital and in the community for personalized treatment in complex chronic patients. The development includes a significant integrative component of self-care management by the patient and / or the primary caregiver.

Following the completion of the technological development, clinical trials will be held in four organizations throughout Europe - Assuta Hospital in Ashdod in cooperation with the Maccabi community in Ashdod, two centers in Catalonia and the Groningen region in the Netherlands. The purpose of the studies is to assess the impact of the implementation of the model, processes and digital tools that will be built during the project.

DETAILED DESCRIPTION:
The intervention in this study consists of two parts:

1. Integrative treatment in the community, which includes a close follow-up with a coordinating nurse for three months after discharge from the hospital.
2. Empowering the patient to self-manage his or her health by using applications for smart devices.

The study protocol:

1. Recruitment of participants during the patient's hospitalization after the patient is identified as a complex patient, explanation of the study and signing the consent form.
2. Evaluation process for the patient, using valid questionnaires, in order to determine the baseline level at the entrance to the study.
3. Distribution of research kit and related accessories and training.
4. Close monitoring for three months in the community after discharge from the hospital and use of the research kit.
5. Reassessment of the patient at the exit of the study.

ELIGIBILITY:
Inclusion Criteria:

* All Maccabi members who arrive at the ER in an unplanned manner
* Age over 65
* Living in a home and not in a nursing home
* LACE> 7
* At least three of the following conditions:

  * Multiple drugs - regular use of four or more drugs
  * More than one case of hospitalization or visit to the ER in the past year
  * Malnutrition
  * Elements of low socio-economic status
* The patient and / or the main caregiver speak Hebrew, English or Russian
* The patient or primary caregiver has a password to the Maccabi Online website
* The patient and / or the primary caregiver have basic technological knowledge in the use of the applications
* The patient has wireless Internet access at home (via Wifi or through a cellular connection)

Exclusion Criteria:

* Patients with cognitive or dementia problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Re-Hospitalizations and emergency room visits in the short term after discharge from the hospital | One month
  Number of hospitalizations and emergency room visits after discharge
Re-Hospitalizations and emergency room visits in the long term after discharge from the hospital | One year
  Number of hospitalizations and emergency room visits after discharge
Length of hospitalization | Less then one month
  In days

SECONDARY OUTCOMES:
Compliance with the assignments in the discharge program guidelines | One year
  At the time of discharge from the hospital, the patient receives a list of tasks to be performed as part of the release letter. We would like to know how many out of this tasks were carried out
Community health services use | One year
  Number of appointments made by the patient during the follow up time for primary physician, professionals, laboratory tests and imaging, physiotherapy and nutritionist.
Evaluation of usability of the technology systems developed | One year
  Using questionnaires for nurses and patients to express their opinion on the use of the technology systems in the project and how much these systems assisted them
Cost-benefits evaluation for the intervention | One year
  Economic evaluation of tests and services saved as a result of active and orderly monitoring of the patient
Assessment of satisfaction of patients from all the projects components (The follow up and the technology systems) | One year
  Using satisfaction questionnaires to be passed at the end of the study
Assessment of satisfaction of medical staff from all the projects components (The follow up and the technology systems) | One year
  Using satisfaction questionnaires to be passed at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bella Azaria, Doctor, Study Director — Assuta Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The European Union's Horizon 2020 Call for Action — https://ec.europa.eu/research/participants/portal/desktop/en/opportunities/h2020/topics/phc-25-2015.html